CLINICAL TRIAL: NCT05758519
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy and Safety of QLS1128 Orally in Symptomatic Participants With Mild to Moderate COVID-19
Brief Title: A Study to Compare QLS1128 With Placebo in Symptomatic Participants With Mild to Moderate COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLS1128-301
Record Dates: First submitted 2023-03-06; First posted 2023-03-07 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLS1128 (Experimental)
  Interventions: Drug: QLS1128
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QLS1128 — QLS1128
  Arms: QLS1128
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 3 Study to Evaluate the Efficacy and Safety of QLS1128 Orally in Symptomatic Participants With Mild to Moderate COVID-19

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between ages of 18-80 years.
2. Confirmed SARS-CoV-2 infection as determined by RT-PCR or antigen test in any specimen collected within 120 hours prior to randomization.
3. Initial onset of the COVID-19-related symptoms/signs within 48 hours prior to the randomization,and any of the following conditions are met on the day of randomization.

   1. Score ≥2 for at least one symptom of body pain or muscle pain, headache,stuffy or runny nose,sore throat,cough,shortness of breath or difficulty breathing.
   2. Risk factors associated with progression to severe/critical COVID-19 with a score ≥1 for at least one symptom of fever,muscle or body pain, headache,stuffy or runny nose,sore throat,cough,shortness of breath or difficulty breathing.
   3. Score ≥1 for fever,with a score ≥1 for at least one symptom of muscle or body pain,headache,stuffy or runny nose,sore throat,cough,shortness of breath or difficulty breathing.

Exclusion Criteria:

1. Previous treatment with QLS1128 sustained-release tablets or other 3CL protease inhibitors failed.
2. has received vaccines within 28 days prior to screening or planned to receive vaccines during the study period (including but not limited to COVID-19 vaccine).
3. Those who have a history of SARS-CoV-2 infection and still have symptoms related to COVID-19 during the screening period.
4. A history of SARS-CoV-2 infection, and the time of diagnosis of the latest infection to the time of diagnosis of the current infection is not more than 28 days.
5. Has received local approved anti-SARS-CoV-2 drugs within 7 days before screening or plan to receive them during the study period.
6. Has received monoclonal antibody against SARS-CoV-2 virus within 1 year prior to screening.
7. Has received convalescent plasma therapy for COVID-19 patients or expect to receive convalescent plasma therapy for COVID-19 patients during the trial.
8. Has received any CYP3A4/2C8 strong inducer within 14 days prior to screening or plan to receive any CYP3A4/2C8 strong inducer during the study period.
9. A known history of active liver disease , including acute/chronic hepatitis B, hepatitis C, cirrhosis, or acute liver failure.
10. Allergic or have contraindications to test drugs or test drug excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2023-03-07 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to sustained recovery of COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when 11 COVID-19 symptoms get scores of 0 for three consecutive days

SECONDARY OUTCOMES:
Viral load | Baseline to Day 4
  Changes of viral load from baseline on Day 4
Time to sustained recovery/ alleviation of each COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when each COVID-19 symptoms get scores of 0 for two consecutive days,or the severity of each COVID-19 symptoms downgrade for two consecutive days
Time to sustained recovery/ alleviation/exacerbation of first COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when first COVID-19 symptoms get scores of 0 for three consecutive days,or the severity of first COVID-19 symptoms downgrade for three consecutive days,or the severity of first COVID-19 symptoms deteriorate for two consecutive days
Time to sustained alleviation of COVID-19 symptoms | Baseline through Day 29
  The time from the start of treatment to the time when the severity of 11 COVID-19 symptoms downgrade for two consecutive days
The time when the virus first turn negative | Baseline through Day 29
  The time when the virus first turn negative
All-cause mortality, COVID-19 related mortality | Baseline through Day 29
  All-cause mortality, COVID-19 related mortality
WHO 11-point ordinal scale | Baseline through Day 29
  Change of WHO 11-point ordinal scale from baseline at different visits
The Adverse events | Baseline through Day 29
  TEAEs associated with drug,SAE associated with drug, adverse events leading to withdrawal, vital signs, physical examination, laboratory examination, 12-lead electrocardiogram, etc

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Pharmaceutical Co., Ltd., Jinan, Shandong, China